CLINICAL TRIAL: NCT03656419
Title: Action of Antimicrobial Photodynamic Therapy With Red Leds in Microorganisms Related to Halitose: Clinical Controlled and Randomized Trial
Brief Title: Photodynamic Therapy With Red Leds in Microorganisms Related to Halitosis
Acronym: halitosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ana Carolina Costa da Mota, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Halitose
Record Dates: First submitted 2018-07-17; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Halitosis
Keywords: Halitosis; Photodynamic Therapy; qPCR
MeSH Terms: conditions — Halitosis | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: A controlled, quantitative cross-sectional clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aPDT group (Experimental): For photodynamic therapy will be used an equipment developed for this project with emission of red LED (660nm) and tip of 2.84 cm² .One session of the Chimiolux® photosensitizing aPDT will be performed, at a concentration of 0.005%, to be applied enough to cover the middle third and back of the tongue for 2 minutes for incubation. Four points will be irradiated with a distance of 1cm between the points, considering the scattering halo and the effectiveness of aPDT. The LED apparatus will be previously calibrated with wavelength 660 nm, with energy of 72 J, power of 800 mW for 90 seconds per point, creep of 282mW / cm².
  Interventions: Procedure: photodynamic therapy
- Tongue Scraper (Active Comparator): Tongue scraper 10 times in the tongue, from the back to the front.
  Interventions: Procedure: Tongue scraper
- aPDT and tongue scraper (Experimental): Tongue scraper 10 times in the tongue, from the back to the front. For aPDT will be used an equipment developed for this project with emission of red LED (660nm) and tip of 2.84 cm² . One session of the Chimiolux® photosensitizing aPDT will be performed, at a concentration of 0.005%, to be applied enough to cover the middle third and back of the tongue for 2 minutes for incubation. Four points will be irradiated with a distance of 1cm between the points. Based on previous studies carried out with the aPDT for the treatment of halitosis the apparatus will be previously calibrated with wavelength 660 nm, with energy of 72 J, power of 800 mW for 90 seconds per point, creep of 282mW / cm².
  Interventions: Procedure: photodynamic therapy; Procedure: Tongue scraper

INTERVENTIONS:
Procedure: photodynamic therapy — aPDT with methylene blue and red led irradiation.
  Arms: aPDT and tongue scraper; aPDT group
Procedure: Tongue scraper — Tongue scraper 10 times from de back to the top.
  Arms: Tongue Scraper; aPDT and tongue scraper

SUMMARY:
Halitosis is the term used to describe any unpleasant odor relative to expired air regardless of its source. The prevalence of halitosis in the population is approximately 30%, of which 80-90% of the cases originate in the oral cavity resulting from proteolytic degradation by gram negative anaerobic bacteria. Antimicrobial photodynamic therapy (aPDT) has been widely used and with very satisfactory results in the health sciences, it involves the use of a non-toxic dye, called photosensitizer (FS), and a light source of a specific wavelength in the presence of the oxygen in the medium. This interaction, is capable of creating toxic species that generate cell death. The advantages of this approach are to avoid resistance to target bacteria and damage to adjacent tissues as the antimicrobial effect is confined only to areas covered by the dye and irradiated by light acting on the target organism rapidly, depending on the dose of light energy and power output. The objective of this controlled clinical study is to verify the effect of aPDT in the treatment of halitosis by evaluating the formation of volatile sulfur compounds with gas chromatography and microbiological analysis before and after treatment. Will be included in this research young adults in the age group between 18 to 25 years with diagnosis of halitosis. The selected subjects will be divided into 3 groups, G1 aPDT, G2 Scraper and G3 aPDT and scraper. All subjects will be submitted to microbiological analysis and evaluation with Oral ChromaTM before, after treatment and followed up of 7, 14 and 30 days For the evaluation of the association of the categorical variables will be used Chi-square test and Fisher's Exact Test, to compare the means will be used tStudent test and Analysis of variance (ANOVA) and to analyze the correlation between the continuous variables will be applied the correlation test by Pearson. In the analyzes of the experimental differences in each group the Wilcoxon test will be used. For all analyzes a level of significance of 95% (p <0.05) will be considered.

DETAILED DESCRIPTION:
The study will follow the regulatory norms of research in humans with favorable opinion of the Research Ethics Committee of the University Nove de Julho number, and the responsible ones of the participants will sign the consent form free after clarifications for authorization of the participation in the research, according to Resolution 466/12 of the National Health Council.

Type of study: A controlled, quantitative cross-sectional clinical study. Hypothesis Null hypothesis: There is no alteration of halitosis after the use of photodynamic therapy employing the use of blue dye and red LED.

There is no microbiological alteration after antimicrobial photodynamic therapy.

Experimental hypothesis: There is a decrease in halitosis after the use of photodynamic therapy using blue dye and red LED associated or not with the tongue scraper.

There is microbiological alteration after antimicrobial photodynamic therapy.

• Research Subjects For this study will be evaluated young adults of both sexes, enrolled regularly in the Dentistry Clinic of the University Nove de Julho - São Paulo.

Inclusion criteria Included in this study are young adults between the ages of 18 and 25, with an informed consent form and authorization for the diagnosis and treatment of halitosis.

Young adults diagnosed with halitosis presenting Oralchroma S2H ≥ 112 ppb and / or CH3SH ≥ 26.

The selected subjects will be divided into 3 groups. There will be 1 session for each group. All samples from the subjects will be submitted to microbiological analysis and evaluation with Oral ChromaTM before and after treatment followed by controls of 7, 14 and 30 days.

Microbiological analysis

Samples of the lingual plaque will be collected using a sterile swab that will be passed on the surface of the tongue back with unique movement and light pressure. Samples will be deposited in sterile tubes that will be identified and stored at -80 ° C until analyzed. After thawing, the samples will be vortexed for one minute. For extraction of the bacterial DNA samples will be boiled for 10 minutes and then centrifuged at 10,000 rpm for 10 minutes. The supernatant will be placed in a new microtube containing 100μL phenol / chloroform / isoamyl alcohol (25: 24: 1), followed by ethanol precipitation. The purified DNA will be resuspended in TE buffer. The levels of P. gingivalis, T. forsythia and T. denticola will be analyzed by quantitative PCR. The quantitative analysis will be performed using real-time PCR using the Step One Plus Real-Time PCR System (Applied Biosystem, Foster City, CA, USA) and fluorescently detected products using the Quantimix Easy SYG Kit (Biotools, Madrid, Spain), following the protocol recommended by the manufacturer. To the reaction 10 l will be used SYBR Green 0.5 ul DNA template, 200 mM of each primer (P. gingivalis CATAGATATCACGAGGAACTCCGA TT and AAACTGTTAGCAACTACCGATGTGG; T.forsythia GGGTGAGTAACGCGTATGTAACCT and ACCCATCCGCAACCAATAAA, T. denticola CGTTCCTGGGCCTTGTACA and TAGCGACTTCAGGTACCCTCG; Universal bacteria CCATGAAGTCGGAATCGCTAG and GCTTGACGGGCGGTGT) in total volume of 20 μl. For the standard curve, reactions containing template DNA 2 to 2X105 copies of the analyzed gene (16S rRNA) will be performed using pTOPO plasmids in which the 16S genes of the 14 different organisms will be cloned. As a negative control will be added sterile milliQ water instead of DNA template. Reactions to 16S rRNA will be performed with initial denaturation at 95 ° C for 2 minutes followed by 36 cycles of 94 ° C for 30 seconds, 55 ° C for 1 minute and 72 ° C for 2 minutes and final extension at 72 ° C for 10 minutes 46. Fluorescence will be detected after each cycle and plotted using Step One Plus Real-Time PCR System software (Applied Biosystem, Foster City, CA, USA). To ensure the specificity of the products detected by fluorescence and to avoid detection of primer dimers, the detection will be performed to a degree below the dissociation temperature of the amplicons. All samples will be analyzed in duplicate and each dilution of the plasmids to the standard curve in triplicate. The purpose of the microbiological evaluation will be to verify the effectiveness of the photodynamic therapy for the treatment of halitosis, complementing the clinical evaluation.

Assessment of halitosis level The air collection will follow the OralChromaTM Manual Instruction, where the participant is instructed to make a mouthwash with cysteine (10 mM) for 1 minute to differentiate the CSV origin and remain mouth closed for 1 minute. A manufacturer's own syringe for collection of mouth air will be introduced into the patient's mouth with the plunger fully inserted. The patient closes his mouth, breathes through his nose and waits with his mouth closed for 1 minute. You will be asked not to touch the tip of the syringe with your tongue. The plunger will be pulled out, re-empties air from the syringe into the patient's mouth and again pulls the plunger to fill the syringe with the breath sample. Clean the tip of the syringe to remove moisture from the saliva, place the gas injection needle in the syringe, adjust the plunger to 0.5 ml. It is injected into the door of the appliance in a single movement.

OralChromaTM allows the capture of gas concentration values by measuring the CSV thresholds (from 0 to 1000 ppb), very accurately after 8 minutes.

The results are stored on the device itself and can be retrieved and viewed at any time for comparison before and after treatment.

From the analysis of CSV captured by the system:

* Sulfide: originates mainly from the bacteria present on the back of the tongue. Values above 112 ppb are indicators of halitosis.
* Methylmercaptan: predominantly higher in the periodontal pockets. Values up to 26 ppb are considered normal. Periodontal disease typically results in a high ratio of methylmercaptan / sulfhydride (> 3: 1)
* Dimethyl sulphide: both may be of periodontal origin or systemic (intestinal, hepatic, pulmonary) origin. It can also be caused, temporarily, by the ingestion of certain foods and beverages. The perception threshold of dimethylsulphide is the lowest, 8 ppb.

To avoid changes in halimetry, the examination will be conducted in the morning and participants will be instructed to follow the following guidelines: 48 hours before the evaluation avoid ingesting food with garlic, onion and strong seasoning, alcohol consumption and use of oral antiseptic. On the day of the evaluation, in the morning, you can eat up to 2 hours before the exam, abstain from coffee, candies, chewing gum, oral hygiene products and perfumed personnel (aftershave, deodorant, perfume, creams and / or tonic) and the brushing will be only with water.

For the photodynamic therapy will be used an equipment developed for this project with emission of red LED (660nm) and tip of 2.84 cm² in diameter.

At the moment of application of the aPDT will be present only the volunteer to be treated and the professional responsible, both using specific eye protection glasses. The active tip of the laser will be coated with clear disposable plastic (PVC) (avoiding cross contamination and hygiene) and the professional will be properly dressed.

One session of the Chimiolux® photosensitizing aPDT will be performed, at a concentration of 0.005% (165μm), to be applied enough to cover the middle third and back of the tongue for 5 minutes for incubation, the excess will be removed with sucker in order to maintain the wet surface with the photosensitizer itself, without the use of water. Four points will be irradiated with a distance of 1cm between the points, considering the scattering halo and the effectiveness of aPDT (figure 5). Based on previous studies carried out with the aPDT for the treatment of halitosis the apparatus will be previously calibrated with wavelength 660 nm, with energy of 72 J, power of 800 mW for groups 1 and 3 that will be irradiated for 90 seconds per point, creep of 282mW / cm².

Organization and Statistical Processing of Data

The data will be tabulated and treated in the program Bioestat 5.0 The descriptive statistics of the data will be performed. For the evaluation of the association of categorical variables, the Chi-square test and Fisher's Exact Test will be used to compare the means will be used Student's t test and Analysis of variance (ANOVA) and to analyze the correlation between the continuous variables will be applied the test of Pearson correlation. In the analyzes of the experimental differences in each group the Wilcoxon test will be used. For all analyzes a level of significance of 95% (p <0.05) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Included in this study are young adults between the ages of 18 and 25, with an informed consent form and authorization for the diagnosis and treatment of halitosis.

Young adults diagnosed with halitosis presenting Oralchroma S2H ≥ 112 ppb and / or CH3SH ≥ 26.

Exclusion Criteria:

* With dentofacial anomalies,
* In orthodontic and / or orthopedic treatment,
* Using a removable device, implant and / or prosthesis,
* With periodontal disease,
* With teeth with carious lesions,
* In cancer treatment,
* On antibiotic treatment up to 1 month prior to the survey,
* Pregnant,
* With hypersensitivity to the photosensitizer to be used.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-10-24 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Results after treatment with gás chromatography | 30 days
  If halitosis reduces in patients after treatment

SECONDARY OUTCOMES:
Microbiological Analysis after treatment with qPCR analisys | 30 days
  If aPDT reduces the microorganism related to halitosis after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Bussadori, PhD, Study Director — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Mota ACC, Goncalves MLL, Horliana ACRT, Deana AM, de Souza Cavalcante LA, Gomes AO, Mayer MPA, Suguimoto ESA, Fernandes KPS, Mesquita-Ferrari RA, Prates RA, Motta LJ, Bussadori SK. Effect of antimicrobial photodynamic therapy with red led and methylene blue on the reduction of halitosis: controlled microbiological clinical trial. Lasers Med Sci. 2022 Mar;37(2):877-886. doi: 10.1007/s10103-021-03325-x. Epub 2021 May 13. PMID 33987732